CLINICAL TRIAL: NCT01969019
Title: A Randomized Trial of Intravenous Pulse Versus Sequential Steroid Therapy for Patients With Graves' Orbitopathy
Brief Title: A Prospective, Randomized Trial of Intravenous Pulse Versus Sequential Steroid Therapy for Patients With Graves' Orbitopathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhu, Attending, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCEMD015
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Graves' Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Methylprednisolone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- methylprednisolone (Active Comparator): intravenous MP: 0.5g weekly for six weeks followed by 0.25g weekly for six weeks
  Interventions: Drug: methylprednisolone, prednisone
- methylprednisolone plus prednisone (Active Comparator): intravenous MP 0.5g daily for three days per week, twice, followed by 0.25g daily for three days per week, twice, and followed by tapering oral prednisone (starting with 60mg/d, then10 mg less/week than each previous week for the next 3 weeks, then20mg/week at the 5th week followed with 5mg less/week than each previous week for the next 3 weeks)
  Interventions: Drug: methylprednisolone, prednisone

INTERVENTIONS:
Drug: methylprednisolone, prednisone

SUMMARY:
This study was designed to compare the efficacy and safety of 4.5g iv MP administered in 12 weeks and 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients should meet the criteria of either a or b and together with c, d and e to include into the study.

  a. Lid retraction with any one of the following: i) Thyroid dysfunction ii) Proptosis iii) Optic nerve involvement iv) Extraocular muscle involvement b. Thyroid dysfunction with any one of the following: i) Proptosis ii) Optic nerve involvement iii) Extraocular muscle involvement c. Exclude cases with such ophthalmological signs caused by other diseases. d. Moderate to severe patients defined by EUGOGO. e. Clinical activity score (CAS)≥3/7 f. Normal function of heart, liver and kidney.

Exclusion Criteria:

* Orbital decompression surgery needed immediately
* History of chronic recurrent or active infection
* History of peptic ulcer
* Patients with a history of chronic liver disease or liver disorders； ALT or AST above 2.5 times upper limit of normal
* History of HIV, hepatitis C or hepatitis B Positive
* Cardiovascular or cerebrovascular disease clinically significant
* Uncontrolled diabetes mellitus
* Use of corticosteroids during 12 weeks before to inclusion period
* Pregnant patient or patient who is planning to become pregnant during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
response rate | 3 months

SECONDARY OUTCOMES:
change of CAS, adverse effects and retreat | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Institute of Endocrine and Metabolic Diseases Department of Endocrine and Metabolic Diseases, Ruijin Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhu W, Ye L, Shen L, Jiao Q, Huang F, Han R, Zhang X, Wang S, Wang W, Ning G. A prospective, randomized trial of intravenous glucocorticoids therapy with different protocols for patients with graves' ophthalmopathy. J Clin Endocrinol Metab. 2014 Jun;99(6):1999-2007. doi: 10.1210/jc.2013-3919. Epub 2014 Feb 28. PMID 24606088